CLINICAL TRIAL: NCT01540513
Title: PET/CT Evaluation of Primary and Metastatic Brain Tumors With a Novel Radioiodinated Phospholipid Ether Analogue I-NM404
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RO11360; 2011-0830 (Other: Institutional Review Board); NCI-2012-02080 (Registry Identifier: NCI Trial ID); A539300 (Other: UW Madison); SMPH\RADIOLOGY\RADIOLOGY (Other: UW Madison)
Record Dates: First submitted 2012-02-14; First posted 2012-02-28 (Estimated); Results first posted 2017-12-11 (Actual); Last update posted 2019-12-02 (Actual); Status verified 2018-02

CONDITIONS: Glioblastoma Multiforme; Brain Metastases
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- I124-NM404 brain metastases or GBM imaging (Experimental): injection of I-124NM404 for imaging
  Interventions: Drug: NM404

INTERVENTIONS:
Drug: NM404 — injection of 5.0mCi I-124 NM404 Arms: I124-NM404 brain metastases or GBM imaging
  Other Names:
  PET imaging with I-124 NM404
Drug: NM404 — injection of an experimental imaging agent, 5mCi I-124NM404

SUMMARY:
The purpose of this study is to evaluate diagnostic imaging techniques using 124I-NM404 PET/CT in human brain tumors. This goal will be accomplished by quantifying tumor uptake and determining the optimal PET/CT protocol, comparing PET tumor uptake to MRI, and calculating tumor dosimetry. The long-term goals of this research are to improve the diagnosis and treatment of malignant brain tumors by using radioiodinated NM404

ELIGIBILITY:
Inclusion Criteria:

* Participants will have a contrast enhanced brain MRI which documents evidence of primary or metastatic brain tumor or suspected tumor recurrence after therapy
* Tumor size at least 1.5 cm in greatest axial dimension on MRI. MRI must be obtained within 2 months of study inclusion
* Adult patients 18 or older
* Female patients must not be pregnant or breast feeding and both women of childbearing potential, and men, must use appropriate means of contraception and must be maintained for at least 45 days after injection of 124I-NM404 Participants must not attempt to become pregnant during this time
* Platelet count must be ≥ 160,000/µl, Hematocrit must be ≥ 22%, Leukocyte count must be ≥ 3,000/µL, Creatinine must be ≤ 2.5 mg/dL, ALT must be ≤ 130 U/L, AST must be ≤ 100 U/L, and urine or serum pregnancy test must be negative for pregnancy
* Patient provides informed consent
* Karnofsky score ≥ 60
* For previously treated brain tumors, targeted brain therapy (radiation or drug) must have concluded ≥2 months prior to injection of 124I-NM404

Exclusion Criteria:

* Life expectancy of < 3 months
* Allergy to potassium iodide (SSKI or Thyroshield)
* Unwilling or unable to complete 3 separate PET/CT imaging sessions of 90 minutes each over 3 days
* Pregnancy or breast-feeding during time of study and/or anticipated breast feeding at any time for 45 days after injection of 124I-NM404.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-03; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lance Hall, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Hospital and Clinics, Madison, Wisconsin, United States

REFERENCES:
- [Result] Hall LT, Titz B, Robins HI, Bednarz BP, Perlman SB, Weichert JP, Kuo JS. PET/CT imaging of the diapeutic alkylphosphocholine analog 124I-CLR1404 in high and low-grade brain tumors. Am J Nucl Med Mol Imaging. 2017 Sep 1;7(4):157-166. eCollection 2017. PMID 28913154
- See also: Impact of PET and MRI threshold-based tumor volume segmentation on patient-specific — http://iopscience.iop.org/article/10.1088/1361-6560/aa716d/meta
- See also: PET/CT imaging of the diapeutic alkylphosphocholine analog 124I-CLR1404 in high and low-grade brain tumors — http://www.ajnmmi.us/files/ajnmmi0058850.pdf
- See also: University of Wisconsin Carbone Cancer Center — https://cancer.wisc.edu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from March 2012 to September 2014 at the University of Wisconsin Hospital and Clinics.
Groups:
- I124-NM404 Brain Metastases or GBM Imaging: Participants injected with 185 MBq ± of 124I-CLR1404 intravenously over a period of 1 to 2 minutes, followed by a flush of 10 mL of normal saline. Subjects returned for PET/CT imaging at 6-, 24-, and 48-hours post-injection.
  Participants received 3 drops of potassium iodide by mouth (1 gm/ml) 1 to 24 hours prior to injection of 124I-CLR1404 and continued additional daily doses prior to each PET/CT scan for 3 consecutive days.
Period: Overall Study
Arm/Group | I124-NM404 Brain Metastases or GBM Imaging
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | I124-NM404 Brain Metastases or GBM Imaging
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 1
Age, Continuous [Mean (Full Range); unit: years] | 43.9 [23 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Tumor to Background Ratios (TBR) Post-imaging for All Lesions With PET Uptake
Description: TBR is calculated by using tumor/lesion SUVmax and dividing by contralateral normal brain background SUVmean value. Imaging performed at 24- and 48 hours post injection.
Time Frame: 24- and 48 hours post injection
Population: Of 12 subjects, only 8 had evaluable data.
Measure: Mean (Standard Deviation); unit: Ratio of PET SUV
Arm/Group | I124-NM404 Brain Metastases or GBM Imaging
Number analyzed (Participants) | 8
Ratio of PET SUV
  24 hours | 8.25 (4.16)
  48 hours | 8.75 (3.60)

2. Primary Outcome: Tumor to Background Ratios (TBR) Post-imaging for Confirmed Malignant Tumors
Description: TBR is calculated by using tumor/lesion SUVmax and dividing by contralateral normal brain background SUVmean value. Imaging performed at 24-, and 48 hours post injection.
Time Frame: 24- and 48 hours post injection
Population: Of 12 participants, 8 had evaluable TBR data.
Measure: Mean (Standard Deviation); unit: Ratio of PET SUV
Arm/Group | I124-NM404 Brain Metastases or GBM Imaging
Number analyzed (Participants) | 8
Ratio of PET SUV
  24 hours | 9.32 (4.33)
  48 hours | 10.04 (3.15)

3. Primary Outcome: Tumor to Blood Pool Ratios Post-imaging for All Lesions With PET Uptake
Description: Tumor to blood pool ratio (tumor SUVmax to superior sinus SUVmean) was calculated at each time point. Tumor to blood pool is calculated by using tumor/lesion SUVmax and dividing by blood pool SUVmean from placing a region of interest in the posterior sagittal sinus near the confluence of sinuses. Imaging performed at 24- and 48 hours post injection.
Time Frame: 24- and 48 hours post injection
Population: Of 12 participants, 8 had evaluable TBR data.
Measure: Mean (Standard Deviation); unit: Ratio of PET SUV
Arm/Group | I124-NM404 Brain Metastases or GBM Imaging
Number analyzed (Participants) | 8
Ratio of PET SUV
  24 hours | 2.86 (1.77)
  48 hours | 2.93 (2.07)

4. Primary Outcome: Tumor to Blood Pool Ratios Post-imaging for Confirmed Malignant Tumors
Description: Tumor to blood pool ratio (tumor SUVmax to superior sinus SUVmean) was calculated at each time point. Tumor to blood pool is calculated by using tumor/lesion SUVmax and dividing by blood pool SUVmean from placing a region of interest in the posterior sagittal sinus near the confluence of sinuses. Imaging performed at 24-, and 48 hours post injection.
Time Frame: 24- and 48 hours post injection
Population: Of 12 participants, 8 had evaluable tumor to blood pool ratio data.
Measure: Mean (Standard Deviation); unit: Ratio of PET SUV
Arm/Group | I124-NM404 Brain Metastases or GBM Imaging
Number analyzed (Participants) | 8
Ratio of PET SUV
  24 hours | 3.35 (1.75)
  48 hours | 3.45 (2.15)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for up to 48 hours (until the time of the final scan).
Description: Subjects are monitored for adverse events (AEs) by the research team and reported by the principle investigator or co-investigators. Subjects are observed during the injection of 124I-NM404 and for 30 minutes after injection. Subjects are also monitored at each PET/CT scanning session. Approximately 2 - 4 weeks after injection of 124I-NM404, subjects were contacted by phone or other means and/or medical records were reviewed, if available, to assess for any AEs. AE data collection is complete.
Arm/Group | I124-NM404 Brain Metastases or GBM Imaging
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes